CLINICAL TRIAL: NCT05743153
Title: OPTIMIZE-UC: Feasibility of a Multimodal Intervention Program to Optimize Treatment Outcomes in Ulcerative Colitis: A Prospective Pilot Study
Brief Title: Feasibility of a Multimodal Intervention Program to Optimize Treatment Outcomes in Ulcerative Colitis
Acronym: OPTIMIZE-UC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 114110
Record Dates: First submitted 2023-01-20; First posted 2023-02-24 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ulcerative colitis (Experimental): Patients participate in multimodal intervention
  Interventions: Behavioral: Multimodal intervention program

INTERVENTIONS:
Behavioral: Multimodal intervention program — Exercise intervention: combined endurance and resistance training three times a week using workout video's which patients can do at home. Advice to exercise at low-intensity for at least 30 minutes per day.
  Nutritional intervention: Patients are advised to aim for optimal energy and protein intake (by registered dietician) and to avoid red meat, processed foods and sweetened drinks. Aiming for a mainly plant based diet.
  Psychological intervention: screening for psychological risk factors and if present, patients are referred to a psychologist for psychological support.

SUMMARY:
This is a prospective, interventional pilot study to assess the feasibility and optimal timing of a multimodal intervention program in Ulcerative Colitis (UC) patients with active disease as well as in patients in remission. Secondly, to demonstrate the effects of a multimodal intervention program on individual patients level and therapy outcomes.

DETAILED DESCRIPTION:
Rationale: Despite considerable advances in the knowledge of UC, and a variation of treatment options, UC still impacts patients' ability to lead a normal life. Clearly, there is an unmet need to improve treatment outcomes. Prehabilitation programs in surgery have shown that the amount of complications is closely related to preoperative physical fitness, nutritional status and psychological well-being. IBD patients often search for self-management strategies to manage their symptoms, however, research focussing on a multimodal intervention approach in parallel to starting new IBD treatment is lacking. Given the potential benefits of intervention programs, limitations of current treatments in terms of improving quality of life and patients' desire for self-management options, we believe that exploring the results of a multimodal intervention program in patients with UC is of high relevance.

Objective/study design: This is a prospective, interventional pilot study to assess the feasibility and optimal timing of a multimodal intervention program in UC patients. Secondly, to demonstrate the effects of a multimodal intervention program on individual patients level and therapy outcomes.

Study population: Patients ≥ 18 years old, with UC. Intervention: Multimodal intervention program including an exercise program, nutritional intervention and psychological evaluation.

Main study parameters/endpoints: This study assesses the feasibility of a multimodal intervention program. Secondary, assesses the effect on:

* Individual patients' level, i.e. physical fitness, nutritional status, mental health, quality of life and work productivity and activity impairment.
* Therapy outcomes, e.g. adherence, number and severity of (S)AEs, corticosteroid use, biochemical and clinical response/remission rates and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Diagnosis of UC confirmed by clinical, endoscopic, and/or histological evidence prior to screening as per standard criteria;
* Ability of subject to participate fully in all aspects of this project;
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Suspicion of differential diagnosis of CD, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis;
* Serious underlying disease other than UC that in the opinion of the investigator may interfere with the subject's ability to participate fully in the study or would compromise subject safety (such as history of malignancies, major neurological disorders, certain orthopedic impairments or any unstable, uncontrolled or severe systemic medical disorder);
* History of alcohol or drug abuse that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures;
* History of psychiatric disorders that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures;
* If female, the subject is pregnant or lactating (< 1 year) or intending to become pregnant;
* Immobilized patients who are not able to complete exercise intervention;
* Illiteracy (disability to read and understand Dutch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Accrural | 24 weeks
  The percentage of approached, eligible participants that are included in the study.
Attrition | 24 weeks
  The percentage of participants who stopped the program prematurely.
Adherence to exercise program | 24 weeks
  Frequency of followed trainings
Adherence to daily exercise goals | 24 weeks
  SQUASH questionnaire
Satisfaction | 24 weeks
  Measured using a patient satisfaction questionnaire
Safety | 24 weeks
  Measured by the number of adverse events occurring during the program

SECONDARY OUTCOMES:
Change in Oxygen Consumption (VO2 max) | 1 year
  Indication of physical fitness
Change in 1 repitition measures | 1 year
  Indication of muscle strength
Change in body weight | 1 year
  Measured in kilograms
Change in fat-free mass | 1 year
  Measured with bioelectrical impedance analysis (BIA)
Change in nutritional status | 1 year
  Measured with Patient Generated Subjective Global Assessment (PG-SGA)
Change in mental health | 1 year
  Hospital Anxiety and Depression scale (HADS questionnaire)
Change in Work Productivity and Activity Impairment | 1 year
  Work Productivity and Activity Impairment Questionnaire (including WPAI-GH)
Change in 36-Item Short Form Health Survey (SF-36) score | 1 year
  Quality of life
Change in EuroQoL (EQ-5D-5L) score | 1 year
  Quality of life
Change in Inflammatory Bowel Disease Questionnaire score | 1 year
  Disease-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Dorien Oomkens, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No